## The GlaxoSmithKline group of companies

| Division | · | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for Study 207674: A randomised, double-blind, parallel group study to evaluate the safety, tolerability and pharmacokinetics of a single dose of GSK2269557 administered via the ELLIPTA <sup>TM</sup> dry powder inhaler to healthy participants. |
|---|---|---|
| <b>Compound Number</b> | : | GSK2269557 |
| <b>Effective Date</b> | : | 08-JUN-2017 |

## **Description:**

The purpose of this reporting and analysis plan (RAP) is to:

• Describe the safety, tolerability, and pharmacokinetics analyses required for the study which will be provided to the study team members to convey the content of the reporting efforts, specifically Statistical Analysis Complete (SAC).

### **Author's Name and Functional Area:**

| PPD | | 10 MAN 2017 |
|--------------------|-------------------------|-------------|
| Manager, Statistic | s (Clinical Statistics) | 19-MAY-2017 |

## Reviewed by:

| PPD | Manager, (Clinical Pharmacology) |
|-----|--------------------------------------------|
| | Programming |
| | Clinical Investigation Lead |
| | Global Clinical Safety & Pharmacovigilance |
| | Safety physician |
| | Medical Writer |
| | Data Manager |
| | Drug Metabolism and Pharmacokinetics |

Approved via e-mail by:

| PPD | • | 07-JUN-2017 |
|-------------|----------------------|-------------|
| Director (C | Clinical Statistics) | U/-JUN-201/ |
| PPD | | 00 HDI 2017 |
| Manager, I | Programming | 08-JUN-2017 |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited

## **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | REPO | RTING & | ANALYSIS PLAN SYNPOSIS | 4 |
| 2. | STIMIN | IARY OF | KEY PROTOCOL INFORMATION | 5 |
| ۷. | 2.1. | | to the Protocol Defined Statistical Analysis Plan | |
| | 2.1. | | | |
| | 2.2. | | esign | |
| | 2.4. | | al Hypotheses | |
| | 2.4. | Statistica | ii i iypotileses | 0 |
| 3. | PLANI | NED ANA | LYSES | <mark>6</mark> |
| | 3.1. | Final Ana | alyses | 6 |
| 4. | ANAL` | YSIS POF | PULATIONS | 6 |
| | 4.1. | | Deviations | |
| 5. | | | ONS FOR DATA ANALYSES AND DATA HANDLING | |
| 5. | | | S | 7 |
| _ | OT LID | V DODLII | ATION ANALYOFO | 0 |
| 6. | | | ATION ANALYSES | |
| | 6.1. | Overviev | v of Planned Analyses | 8 |
| 7. | PRIMA | | FISTICAL ANALYSES | |
| | 7.1. | Pharmac | cokinetic Analyses | |
| | | 7.1.1. | Overview of Planned Pharmacokinetic Analyses | |
| | | 7.1.2. | Drug Concentration Measures | |
| | | 7.1.3. | Pharmacokinetic Parameters | |
| | | | 7.1.3.1. Deriving Pharmacokinetic Parameters | 9 |
| | | | 7.1.3.2. Statistical Analysis of Pharmacokinetic | |
| | | | Parameters | 11 |
| 8. | SECO | NDARY S | STATISTICAL ANALYSES | 11 |
| | 8.1. | | nalyses | |
| | | 8.1.1. | Overview of Planned Safety Analyses | |
| | | | 8.1.1.1. Statistical Analysis of Safety Parameters | |
| ^ | DEEE | DENOCO | | |
| 9. | KEFE | RENCES. | | 13 |
| 10. | APPE | NDICES | | 14 |
| | 10.1. | Appendix | x 1: Time & Events | 15 |
| | | 10.1.1. | Protocol Defined Time & Events | 15 |
| | 10.2. | Appendix | x 2: Treatment States and Phases | 20 |
| | | 10.2.1. | Treatment Phases | 20 |
| | | 10.2.2. | Treatment States | 20 |
| | | | 10.2.2.1. Treatment States for AE Data | |
| | 10.3. | Appendix | x 3: Data Display Standards & Handling Conventions | 21 |
| | | 10.3.1. | Study Treatment & Sub-group Display Descriptors | 21 |
| | | 10.3.2. | Baseline Definition & Derivations | 21 |
| | | | 10.3.2.1. Baseline Definitions | <mark>21</mark> |

## CONFIDENTIAL

| | | 10.3.2.2. Derivations and Handling of Missing Baseline | |
|---|---|---|---|
| | | Data | 21 |
| | 10.3.3. | Reporting Process & Standards | 21 |
| 10.4. | Appendi | x 4: Derived and Transformed Data | 24 |
| | 10.4.1. | General | 24 |
| | 10.4.2. | Study Population | 24 |
| | 10.4.3. | J | |
| 10.5. | Appendi | x 5: Premature Withdrawals & Handling of Missing Data | 26 |
| | 10.5.1. | Premature Withdrawals | 26 |
| | 10.5.2. | Handling of Missing Data | 26 |
| | | 10.5.2.1. Handling of Missing Dates | 26 |
| | | 10.5.2.2. Handling of Partial Dates | 27 |
| 10.6. | Appendi | x 6: Values of Potential Clinical Importance | 28 |
| | 10.6.1. | Laboratory Values | 28 |
| | 10.6.2. | ECG | |
| | 10.6.3. | Vital Signs | 29 |
| 10.7. | Appendi | x 7 - Abbreviations & Trade Marks | 30 |
| | 10.7.1. | Abbreviations | 30 |
| | | Trademarks | |
| 10.8. | | x 8: List of Data Displays | |
| | 10.8.1. | 3 | |
| | 10.8.2. | Deliverable [Priority] | |
| | 10.8.3. | Study Population Tables | |
| | 10.8.4. | Safety Tables | |
| | 10.8.5. | Pharmacokinetic Tables | |
| | 10.8.6. | Pharmacokinetic Figures | |
| | 10.8.7. | ICH Listings | 38 |

# 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the Reporting and Analysis Plan |
|---|---|
| Purpose | The purpose of this reporting and analysis plan (RAP) is to describe: |
| | Planned analyses and output for the study. |
| Protocol | <ul> <li>Reporting and Analysis Plan is based on original protocol (Dated: 04-APR-2017) for<br/>study</li> <li>GSK2269557/207674 [GlaxoSmithKline Document Number: 2017N316562_00].</li> </ul> |
| Drimonni | |
| Primary Objective / Endpoint | <ul> <li>Primary objective is to assess the pharmacokinetic profile of a single dose of<br/>GSK2269557 administered via the ELLIPTA™ dry powder inhaler to healthy participants<br/>by derived pharmacokinetic parameters including:</li> </ul> |
| | Area under the plasma drug concentration versus time curve from zero to time t AUC(0-t), Area under the plasma drug concentration versus time curve from zero to 24 hours AUC(0-24), Area under the plasma drug concentration versus time curve from zero to infinity AUC(0-inf∞), Maximum observed plasma drug concentration (Cmax), Time to maximum observed plasma drug concentration (Tmax), Concentration at trough (Ctrough), Terminal half-life (T1/2), where data allow. |
| Study | Randomised, double-blind, parallel group, single dose study in healthy participants. |
| Design | <ul> <li>Approximately 12 participants will be randomised to receive a single dose of<br/>GSK2269557 750 μg or a single dose of GSK2269557 500 μg in a 1:1 ratio.</li> </ul> |
| Analysis<br>Population | Primary: Pharmacokinetic Population (Comprised of All randomised participants who take at least 1 dose of study treatment and for whom a pharmacokinetic sample was obtained and analysed. Participants will be analysed according to the treatment they received). |
| Hypothesis | There are no formal hypotheses being tested in the study; instead an estimation and inference approach will be adopted to evaluate the objectives. |
| Primary<br>Analyses | Pharmacokinetic data will be presented in tabular and/or graphical format and summarized descriptively according to GSK's Integrated Data Standards Library (IDSL) standards. Individual GSK2269557 plasma concentration-time profiles (by treatment and subject) and median/mean (±SD) profiles by treatment group will be plotted and listed. Plasma concentration time data for GSK2269557 will be analyzed by non-compartmental methods using WinNonlin and derived PK parameters summarised and listed. No formal statistical analyses will be conducted. |
| Secondary<br>Analyses | Safety data will be presented in tabular format and summarized descriptively. |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol [Dated: 04-APR-2017].

## 2.2. Study Objective(s) and Endpoint(s)

| Obj | ectives | Endpoints |
|---|---|---|
| Prir | mary (Pharmacokinetic) | Primary (Pharmacokinetic) |
| • | To assess the pharmacokinetic profile of a single dose of GSK2269557 administered via the ELLIPTA dry powder inhaler to healthy participants. | • GSK2269557 plasma concentration data and derived pharmacokinetic parameters including area under the plasma drug concentration versus time curve from zero to time t (AUC(0-t)), area under the plasma drug concentration versus time curve from zero to 24 hours (AUC(0-24)), area under the plasma drug concentration versus time curve from zero to infinity (AUC(0-inf∞)), maximum observed plasma drug concentration (Cmax), time to maximum observed plasma drug concentration (Tmax), Concentration at trough (Ctrough), terminal half-life (T1/2), where data allow. |
| Secondary Objectives (Safety) | | Secondary Endpoints (Safety) |
| • | To assess the safety and tolerability of a single dose of GSK2269557 administered via the ELLIPTA dry powder inhaler to healthy participants. | <ul> <li>Safety and tolerability of GSK2269557 as assessed by clinical monitoring of:</li> <li>Vital Signs</li> <li>Electrocardiogram (ECG)</li> <li>Spirometry</li> <li>Laboratory safety data</li> <li>Adverse events (AEs)</li> </ul> |

## 2.3. Study Design

| Overview of | Overview of Study Design and Key Features |
|---|---|
| Pesign Features Randomised, double-blind, parallel group single centre study to investigate the safety, tolerability, and pharmacokinetics of a single dose of GSK2269557 administered via the ELLIPTAT dry powder inhaler to healthy participants. | |
| Dosing | Patients dosed within 28 days of screening. |
| J | <ul> <li>Study treatment will be administrated on Day 1. Participants will be discharged<br/>after completion of all 24h post dose assessments on Day 2 and if there are no<br/>safety concerns</li> </ul> |
| Treatment<br>Assignment | <ul> <li>Approximately 12 participants will be randomised to receive a single dose of<br/>GSK2269557 750 μg or a single dose of GSK2269557 500 μg in a 1:1 ratio.</li> </ul> |

## 2.4. Statistical Hypotheses

There are no formal hypotheses being tested in the study; instead an estimation and inference approach will be adopted to evaluate the objectives.

## 3. PLANNED ANALYSES

## 3.1. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- [1] All subjects have completed the study as defined in the protocol.
- [2] All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- [3] All criteria for unblinding the randomisation codes have been met.
- [4] Randomisation codes have been distributed according to RandAll NG procedures.

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Endpoint(s) Evaluated |
|---|---|---|
| All Participants<br>Enrolled (APE)<br>Population | <ul> <li>All participants for whom a record exists<br/>on the study database; includes both<br/>screen participants and participants who<br/>are not screened but sign the informed<br/>consent form</li> </ul> | Study Population |
| Safety | All randomised participants who receive at least one dose of study treatment. Participants will be analysed according to the treatment they actually received. | <ul><li>Study Population</li><li>Safety</li></ul> |

| Population | Definition / Criteria | Endpoint(s) Evaluated |
|---|---|---|
| Pharmacokinetic | All randomised participants in the Safety population and for whom a pharmacokinetic sample was obtained and analysed. | • PK |

#### NOTES:

Please refer to Appendix 7 which details the population to be used for each display being generated.

#### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---------|--------------------------------------------------------------|
| 10.1 | Appendix 1: Time & Events |
| 10.2 | Appendix 2: Treatment States and Phases |
| 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| 10.4 | Appendix 4: Derived and Transformed Data |
| 10.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| 10.6 | Appendix 6: Values of Potential Clinical Importance |

## 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Analyses

The study population analyses will be based on the "Safety" or "APE" population, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 8: List of Data Displays.

 Table 2
 Overview of Planned Study Population Analyses

| Display Type | Data I | Display's Gen | erated |
|---|---|---|---|
| | Figure | Table | Listing |
| Randomisation | | | |
| Randomisation | | | Y |
| Subject Disposition | | | |
| Subject Disposition | | Υ | |
| Reasons for Screening Failures | | Υ | Υ |
| Reasons for Withdrawals | | | Y |
| Important Protocol Deviations | | Υ | Y |
| Inclusion and Exclusion Criteria Deviations | | | Y |
| Demography | | | |
| Demographics Characteristics | | Υ | Y |
| Age Ranges | | Υ | |
| Race & Racial Combinations | | Υ | Y |
| Study Populations | | Υ | |
| Medical Condition & Concomitant Medications | | | |
| Medical Conditions (Current/Past) | | | Y |
| Concomitant Medication | | | Y |

#### NOTES:

• Y = Yes display generated.

## 7. PRIMARY STATISTICAL ANALYSES

## 7.1. Pharmacokinetic Analyses

The primary pharmacokinetic analyses will be based on the "Pharmacokinetic" population, unless otherwise specified.

## 7.1.1. Overview of Planned Pharmacokinetic Analyses

Table 3 provides an overview of the planned pharmacokinetic analyses with full details of data displays being presented in Appendix 8: List of Data Displays.

 Table 3
 Overview of Planned Pharmacokinetic Analyses

| Endpoints | Untransformed | | | | Log-Transformed | | | |
|---|---|---|---|---|---|---|---|---|
| | Sum | Summary | | Individual | | Summary | | Individual |
| | F | Т | F | L | F | T | F | L |
| Plasma Concentrations | Y | Υ | Υ | Υ | Υ | Υ | Υ | |
| Derived PK Parameters | | Υ | | Y | | Υ | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 7.1.2. Drug Concentration Measures

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 10.3.3 Reporting Process & Standards).

#### 7.1.3. Pharmacokinetic Parameters

## 7.1.3.1. Deriving Pharmacokinetic Parameters

- Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 10.3.3 Reporting Process & Standards).
- The pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using Win Nonlin Pro.
- All calculations of non-compartmental parameters will be based on actual sampling times recorded during the study.
- Pharmacokinetic parameters described in Table 4 will be determined from plasma GSK2269557 concentration-time data, as data permits.

 Table 4
 Derived Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (C(t)) will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| AUC(0-24) | Area under the concentration-time curve will be calculated to fixed nominal time 24 hours after administration (AUC(0-24)), using the combination of linear and logarithmic trapezoidal methods (i.e., Linear Up/Log Down calculation method in Phoenix WinNonlin Professional). |
| | If a sampling time deviation occurred at nominal time 24 hours after administration (and 24 < t), AUC(0-24) will be calculated using the concentration at time 24 hours after administration post-dose estimated by the method of interpolation. |
| | If nominal time 24 hours after administration > t (or if the concentration at time 24 hours after administration was below then limit of quantification), then the concentration (y) at time 24 hours after administration is estimated using lambda_z and last observed Ct according to the formula: |
| | y=Ct(obser) x e-lambda_z(24-t) |
| | Then the following equation will be used to calculate (AUC(0-24)) where t is the time of last quantifiable plasma concentration. |
| | AUC(0-24) = AUC(0-t) + AUC(t-24) |
| | If lambda_z is not estimable, a partial AUC is not calculated (when 24 > t). |
| AUC(0-<br>inf∞) | Area under the concentration-time curve from zero time (pre-dose) extrapolated to infinite time (AUC(0-inf)) will be calculated as follows: |
| | $AUC(0-inf) = AUC(0-t) + Ct / lambda_z.$ |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| Ctrough | Trough observed concentration, will be obtained directly from the concentration-time data. |
| t½ | Apparent terminal half-life will be calculated as: |
| | $t^{1/2} = \ln 2 / \lambda z$ |
| | (NOTE: λz is the terminal phase rate constant). |

## NOTES:

Additional parameters may be included as required.

## 7.1.3.2. Statistical Analysis of Pharmacokinetic Parameters

There are no planned statistical analyses.

## 8. SECONDARY STATISTICAL ANALYSES

## 8.1. Safety Analyses

## 8.1.1. Overview of Planned Safety Analyses

The safety analyses will be based on the "Safety" population, unless otherwise specified.

Table 5 provides an overview of the planned analyses, with full details being presented in Appendix 8: List of Data Displays.

Table 5 Overview of Planned Safety Analyses

| Endpoint | | Abso | olute | | C | Change from Baselii | | |
|---|---|---|---|---|---|---|---|---|
| | Summary | | Indiv | Individual | | Summary | | ridual |
| | T | F | F | L | T | F | F | L |
| Adverse Events | | | | | | | | |
| All AE's | Υ | | | Υ | | | | |
| All Drug-Related AE's | Υ | | | | | | | |
| Serious AE's | Υ | | | Υ | | | | |
| Non Serious AE's | Υ | | | | | | | |
| Withdrawal AE's | Υ | | | Υ | | | | |
| Laboratory Values | | | | | | | | |
| Clinical Chemistry | | | | | Υ | | | |
| Hematology | | | | | Υ | | | |
| Urinalysis | Υ | | | | | | | |
| ECG's | | | | | | | | |
| ECG Findings | Υ | | | | | | | |
| ECG Values | Υ | | | | Υ | | | |
| Vital Signs | | | | | | | | |
| Vitals Values | | | | | Υ | | | |
| Emergent Vital Signs | | | | Υ | Υ | | | |
| Spirometry | | | | | | | | |
| FEV1 | Υ | | | Υ | Υ | | | |
| FVC | Υ | | | Υ | Υ | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

# 8.1.1.1. Statistical Analysis of Safety Parameters

There are no planned statistical analyses.

## 9. REFERENCES

GlaxoSmithKline Document Numbers 2017N316562\_00 (Original 04-APR-2017): A randomised, double-blind, parallel group study to evaluate the safety, tolerability and pharmacokinetics of a single dose of GSK2269557 administered via the ELLIPTA dry powder inhaler to healthy participants).

## 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 5 | General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.1 | Appendix 1: Time and Events |
| Section 10.2 | Appendix 2: Treatment States & Phases |
| Section 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.4 | Appendix 4: Derived and Transformed Data |
| | General |
| | Study Population |
| | • Safety |
| Section 10.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| Section 10.6 | Appendix 6: Values of Potential Clinical Importance |
| | Laboratory Values |
| | • ECG |
| | Vital Signs |
| Other RAP App | endices |
| Section 10.7 | Appendix 7: Abbreviations & Trade Marks |
| Section 10.8 | Appendix 8: List of Data Displays |

# 10.1. Appendix 1: Time & Events

## 10.1.1. Protocol Defined Time & Events

| | Screening | | Treat | tment Period [ | | | Notes | |
|---|---|---|---|---|---|---|---|---|
| Procedure | (up to 28<br>days<br>before Day<br>1) | <b>-</b> 1 | 1 | 2 | 3 | 6 | Follow-up<br>(10-12 days post dose) | |
| Informed consent | Х | | | | | | | |
| Inclusion and exclusion criteria | X | | | | | | | Recheck clinical<br>status before<br>randomization |
| Demography | Х | | | | | | | |
| Full physical examination including height and weight | Х | | | | | | | |
| Medical history (includes substance usage and current medical conditions) | X | | | | | | | Substances:<br>Drugs, Alcohol,<br>tobacco and<br>caffeine |
| Urine pregnancy test (WOCBP only) | Х | Х | | | | | | |

| | Screening | | Trea | tment Period [ | | | Notes | |
|---|---|---|---|---|---|---|---|---|
| Procedure | (up to 28<br>days<br>before Day<br>1) | -1 | 1 | 2 | 3 | 6 | Follow-up<br>(10-12 days post dose) | |
| HIV, Hepatitis B and C screening | X | | | | | | | If test otherwise performed within 3 months prior to first dose of study treatment, testing at screening is not required |
| Admission to unit | | Х | | | | | | |
| Outpatient visit | | | | | Х | Х | | |
| Discharge | | | | Х | | | | |
| Laboratory assessments (include liver chemistries) | Х | Х | | Х | | | | |
| Urine Drug, Alcohol and Smoking breath test | Х | Х | | | | | | |

| | Screening | | Treat | ment Period [l | Days] | | | Notes |
|---|---|---|---|---|---|---|---|---|
| Procedure | (up to 28<br>days<br>before Day<br>1) | <b>-1</b> | 1 | 2 | 3 | 6 | Follow-up<br>(10-12 days post dose) | |
| | | | | | | | | Screening only:<br>ECG in triplicate |
| 12-lead ECG | X | | Х | X | | | | Day 1: pre-dose, 5 mins & 6 hrs post-dose |
| | | | | | | | | Day 2: before discharge |
| | | | | | | | | Screening only: VS in triplicate |
| Vital signs | Х | | X | X | | | | Day1: pre-dose, 1h and 6h post-dose |
| FEV1 and FVC (triplicate) | Х | | Х | | | | | Day 1: pre-dose,<br>30 min post-dose |
| Brief physical examination | | Х | | | | | | |

| | Screening | | Trea | tment Period [ | Days] | | | Notes |
|---|---|---|---|---|---|---|---|---|
| Procedure | (up to 28<br>days<br>before Day<br>1) | -1 | 1 | 2 | 3 | 6 | Follow-up<br>(10-12 days post dose) | |
| Inhaler training | | X | | | | | | Training conducted by reviewing the Patient Information Leaflet with the participant. Additional training may be conducted at the discretion of the investigator. |
| Dosing study treatment | | | X | | | | | |
| AE review | | | <b>←====</b> | ======== | ======== | ======== | | |
| SAE review | • | _======= | -======= | ======== | ======== | ======= | =====→ | |
| Concomitant medication review | | | Х | Х | Х | Х | X | |
| Pharmacokinetic blood sample | | | X | X | Х | Х | | Day 1: pre-dose, 5 min and 0.5, 2, 6 and 12 hours post-dose. Day 2: 24 hours post-dose. Day 3: 48 hours post-dose Day 6: 120 hours post dose. |

- The timing and number of planned study assessments, including safety and pharmacokinetic assessments may be altered during the course of the study based on newly available data (e.g., for safety purposes or to obtain data closer to the time of peak plasma concentrations) to ensure appropriate monitoring.
- Any changes in the timing or addition of time points for any planned study assessments must be documented and approved by the relevant study team member and then archived in the sponsor and site study files, but will not constitute a protocol amendment. The IRB/IEC will be informed of any safety issues that require alteration of the safety monitoring scheme or amendment of the ICF

## 10.2. Appendix 2: Treatment States and Phases

#### 10.2.1. Treatment Phases

Assessments and events will be classified according to the time of occurrence relative to dosing.

| Treatment Phase | Definition |
|---|---|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start date < Date ≤ Study Treatment Stop Date |
| Post-Treatment | Date > Study Treatment Stop Date |

### 10.2.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment.

#### 10.2.2.1. Treatment States for AE Data

| Treatment<br>State | Definition |
|---|---|
| Pre-Treatment | AE Start Date < Study Treatment Start Date |
| On-Treatment | If AE onset date is on or after treatment start date & on or before the treatment stop date |
| On-Treatment | Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date [+ 1] |
| Post-Treatment | If AE onset date is after the treatment stop date |
| Post-meatinent | AE Start Date > Study Treatment Stop Date |
| Onset Time | If Treatment Start Date > AE Onset Date = AE Onset Date - Treatment Start Date |
| Since First Dose | If Treatment Start Date ≤ AE Onset Date = AE Onset Date - Treatment Start Date +1 |
| (Days) | Missing otherwise |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on eCRF OR value is missing |

#### NOTES:

• If the study treatment stop date is missing then the AE will be considered to be On-Treatment.

# 10.3. Appendix 3: Data Display Standards & Handling Conventions

## 10.3.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| | RandAll NG Data Displays for Reporting | | |
| Code Description | | Description | Order [1] |
| Α | GSK2269557 500 mcg | GSK2269557 500 mcg | 1 |
| В | GSK2269557 750 mcg | GSK2269557 750 mcg | 2 |

#### NOTES:

#### 10.3.2. Baseline Definition & Derivations

#### 10.3.2.1. Baseline Definitions

For all endpoints the baseline value will be the latest pre-dose assessment.

### 10.3.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|----------------------|------------------------------------|
| Change from Baseline | = Post-Dose Visit Value – Baseline |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 10.3.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

## 10.3.3. Reporting Process & Standards

| Troporting Frodood & Ottainaardo | |
|---|---|
| Reporting Process | Reporting Process |
| Software | Software |
| The currently s | upported versions of SAS software will be used. |
| Reporting Area | |
| HARP Server | : uk1salx00175 |
| HARP Area | : \arprod\gsk2269557\mid207674\final_01 |
| QC Spreadsheet | QC Spreadsheet : \ARWORK\gsk2269557\ mid207674\Final_01\Documents |
| Analysis Datasets | |
| Analysis datasets will be created according to CDISC standards | |
| Generation of RTF Files | |
| RTF files for tables will be generated. | |

<sup>1.</sup> Order in which treatments are to be presented in Tables, Figures and Listings.

#### Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - o 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables and figures:
  - Planned time relative to dosing will be used in figures and summaries and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings.
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures and summaries.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Continuous Data Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Reporting of Pharmacokinetic Concentration Data | |
| Descriptive Summary | Refer to IDSL Statistical Principle 6.06.1 |
| Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |
| Reporting of Pharmacokinetic Parameters | |
| Descriptive Summary N, n, geometric mean, 95% CI of geometric mean, standard deviation | |

| Reporting Standards | |
|---|---|
| Statistics.<br>(Log Transformed) | (SD) of logged data and between geometric coefficient of variation (CVb (%)) will be reported. |
| | CVb (%) = $\sqrt{(\exp(SD2) - 1) * 100}$ [NOTE: SD = SD of log transformed data] |
| Parameters Not Being Log Transformed | tmax, first point, last point and number of points used in the determination of Lambda_z. |
| Parameters Not Being<br>Summarised | Additionally include tmax, first point, last point and number of points used in the determination of Lambda_z. |
| Listings | Include the first point, last point and number of points used in the determination of Lambda_z. |
| Graphical Displays | |
| Refer to IDSL Statistical Principles 7.01 to 7.13. | |

## 10.4. Appendix 4: Derived and Transformed Data

#### 10.4.1. General

## **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

### **FEV1 and FVC measurements**

 FEV1 and FVC measurements are to be taken in triplicate, the maximum of the values entered at one time point will be used for the summaries and listings of FEV1 and FVC

### Study Day

- Calculated as the number of days from randomisation date :
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Randomisation Date → Study Day = Ref Date Randomisation Date</li>
  - Ref Data ≥ Randomisation Date → Study Day = Ref Date (Randomisation Date) + 1

## 10.4.2. Study Population

#### **Demographics**

#### Age

- GSK standard algorithms will be used for calculating age where birth date is imputed as:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

## **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>

#### **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula:
  - Duration of Exposure in Days = Treatment Stop Date (Treatment Start Date) + 1
- Subjects who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.

## 10.4.3. Safety

## **ECG Parameters**

#### **RR Interval**

• IF RR interval (msec) is not provided directly, then RR can be derived as :

[1] If QTcB is machine read & QTcF is not provided, then :

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^{3} \right] * 1000$$

 If ECGs are manually read, the RR value preceding the measurement QT interval should be collected values THEN do not derive.

## **Corrected QT Intervals**

 When not entered directly in the eCRF, corrected QT intervals using Bazett's (QTcB) and Fridericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.

• IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

#### **Adverse Events**

MedDRA version 20.0 will be used for coding of AE's.

# 10.5. Appendix 5: Premature Withdrawals & Handling of Missing Data

## 10.5.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion is defined as subjects who receive study treatment and complete all post dose assessments, including the Follow Up Phone Call. |
| | Withdrawn subjects maybe replaced in the study. |
| | All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |

## 10.5.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument : |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing<br/>displays. Unless all data for a specific visit are missing in which case the<br/>data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to<br/>be missing data and should be displayed as such.</li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 10.5.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: |
| | Missing Start Day: First of the month will be used unless this is before the start date of investigational product; in this case the study treatment start date will be used (and hence the event is considered On-treatment as per Appendix 3: Treatment States and Phases). |
| | Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will |

| Element | Reporting Detail |
|---|---|
| | be used. |
| | <ul> <li>Completely missing start or end dates will remain missing, with no imputation<br/>applied. Consequently, time to onset and duration of such events will be<br/>missing.</li> </ul> |
| | Start or end dates which are completely missing (i.e. no year specified) will remain missing, with no imputation applied. |

# 10.5.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant Medications | Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will<br/>be used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day<br/>(dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |
| Adverse<br>Events | Any partial dates for adverse events will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will<br/>be used for the month.</li> </ul> |
| | <ul> <li>However, if these results in a date prior to Week 1 Day 1 and the event<br/>could possibly have occurred during treatment from the partial information,<br/>then the Week 1 Day 1 date will be assumed to be the start date.</li> </ul> |
| | The AE will then be considered to start on-treatment (worst case). |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day<br/>(dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |

# 10.6. Appendix 6: Values of Potential Clinical Importance

## 10.6.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | ↓0.075 | |
| | g/L | Male | | 180 |
| Hemoglobin | | Female | | 180 |
| | | $\Delta$ from BL | ↓25 | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| - | | | Low Flag (< x) | High Flag (>x) |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | mmol/L | $\Delta$ from BL | | ↑ 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

## 10.6.2. ECG

| ECG Parameter | Units | Clinical Concern Range |
|---------------|-------|------------------------|
| | | Lower Upper |
| Absolute | | |

| ECG Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute QTc Interval | msec | > 450 | |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | Change from Baseline | | |
| Increase from Baseline QTc | msec | ≥ 60 | |
| increase from baseline Q10 | msec | > 30 | ≤ 59 |

# 10.6.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

# 10.7. Appendix 7 - Abbreviations & Trade Marks

## 10.7.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AE | Adverse Event |
| APE | All Participants Enrolled |
| AUC(0-24) | Area Under the Plasma Drug Concentration versus Time Curve |
| , , , | from zero to 24 hours |
| AUC(0-∞) | Area under the concentration-time curve from time zero (pre-dose) |
| , , | extrapolated to infinite time |
| AUC(0-t) | Area under the concentration-time curve from time zero (pre-dose) to |
| | last time of quantifiable concentration within a subject across all |
| | treatments |
| BMI | Body mass index |
| CI | Confidence Interval |
| Cmax | Maximum observed concentration |
| Ctrough | Concentration at trough |
| CV | Coefficient of variance |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| FEV1 | Forced expiratory volume in 1 second |
| FVC | Forced Vital Capacity |
| GSK | GlaxoSmithKline |
| hrs | Hours |
| IDSL | Integrated Data Standards Library |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mcg | Micrograms |
| msec | Milliseconds |
| NQ | Non Quantifiable |
| PK | Pharmacokinetic |
| QTc | Corrected QT interval |
| RAP | Reporting and Analysis Plan |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event(s) |
| SAS | Statistical Analysis Software |
| SD | Standard Deviation |
| T1/2 | Terminal Half-life |
| Tmax | Time to maximum observed plasma drug concentration |
| WOCBP | Women of Child Bearing Potential |

## 10.7.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| ELLIPTA |
| HARP |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |
| WinNonlin |

# 10.8. Appendix 8: List of Data Displays

## 10.8.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-----------------------|---------|
| Study Population | 1.1 to 1.8 | N/A |
| Safety | 2.1 to 2.17 | N/A |
| Pharmacokinetic | 3.1 to 3.4 3.1 to 3.2 | |
| Section | Listings | |
| ICH Listings | 1 to 28 | |
| Other Listings | N/A | |

# 10.8.2. Deliverable [Priority]

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------|
| SAC [1] | Statistical Analysis Complete |

#### NOTES:

<sup>1.</sup> Indicates priority (i.e. order) in which displays will be generated for the reporting effort.

# 10.8.3. Study Population Tables

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1 | Safety | ES1 | Summary of Subject Disposition | | SAC [1] |
| 1.2 | APE | ES6 | Summary of Reasons for Screening Failure | | SAC [1] |
| 1.3 | Safety | DV1 | Summary of Important Protocol Deviations | | SAC [1] |
| Demog | raphics | | | | |
| 1.4 | Safety | SP1 | Summary of Study Populations | | SAC [1] |
| 1.5 | Safety | DM1 | Summary of Demographic Characteristics | | SAC [1] |
| 1.6 | Safety | DM11 | Summary of Age Ranges | | SAC [1] |
| 1.7 | Safety | DM5 | Summary of Race and Racial Combinations | | SAC [1] |

# 10.8.4. Safety Tables

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | se Events | | | | |
| 2.1 | Safety | CP_AE1p | Summary of All Adverse Events | | SAC [1] |
| 2.2 | Safety | CP_AE1p | Summary of All Drug-Related Adverse Events | Include total column. | SAC [1] |
| 2.3 | Safety | CP_AE1p | Summary of Serious Adverse Events | | SAC [1] |
| 2.4 | Safety | AE15 | Summary of Common (>=5%) Non-serious Adverse<br>Events by System Organ Class and Preferred Term<br>(Number of Subjects and Occurrences) | | SAC [1] |
| 2.5 | Safety | CP_AE1p | Summary of Adverse Events Leading to Permanent Discontinuation of Study Drug or Withdrawal from Study | | SAC [1] |
| Labs | | | | | 1 |
| 2.6 | Safety | LB1 | Summary of Chemistry Changes from Baseline | | SAC [1] |
| 2.7 | Safety | LB17 | Summary of Emergent Chemistry Results by Potential Clinical Importance (PCI) Criteria | | SAC [1] |
| 2.8 | Safety | LB1 | Summary of Haematology Changes from Baseline | | SAC [1] |
| 2.9 | Safety | LB17 | Summary of Emergent Haematology Results by Potential Clinical Importance (PCI) Criteria | | SAC [1] |

| Safety | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.10 | Safety | UR3b (LB1) | Summary of Urinalysis Results by Planned Timepoint | Use shell UR3b for: pH, glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase as these are collected by dipstick | SAC [1] |
| | | | | Use shell LB1 for: Specific gravity | |
| ECGs | | | | | |
| 2.11 | Safety | EG1 | Summary of ECG Findings | | SAC [1] |
| 2.12 | Safety | EG2 | Summary of ECG Values | | SAC [1] |
| 2.13 | Safety | EG2 | Summary of Change from Baseline in ECG Values | | SAC [1] |
| Vital Si | gns | | | | |
| 2.14 | Safety | VS1 | Summary of Change from Baseline in Vital Signs | | SAC [1] |
| 2.15 | Safety | VS7 | Summary of Emergent Vital Signs Results by Potential Clinical Importance (PCI) Criteria | | SAC [1] |
| Spiron | netry | | | | |
| 2.16 | Safety | | Summary of Spirometry (FVC and FEV1) | See example:<br>uk1salx00175/gsk2269557/mid205759/final/<br>Table 2.35 | SAC [1] |
| 2.17 | Safety | | Summary of Change from Baseline in Spirometry (FVC and FEV1) | See example:<br>uk1salx00175/gsk2269557/mid205759/final/<br>Table 2.38 | SAC [1] |

## 10.8.5. Pharmacokinetic Tables

| Pharma | Pharmacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Cor | PK Concentration Data | | | | |
| 3.1 | PK | PK01 | Summary of Plasma GSK2269557 Pharmacokinetic Concentration-Time Data | | SAC [1] |
| 3.2 | PK | PK01 | Summary of Plasma GSK2269557 Pharmacokinetic Concentration-Time Data (log transformed) | | SAC [1] |
| PK Der | PK Derived Parameters | | | | |
| 3.3 | PK | PK03 | Summary of Derived Plasma GSK2269557<br>Pharmacokinetic Parameters | Parameters with units | SAC [1] |
| 3.4 | PK | PK05 | Summary of Log-Transformed Derived Plasma<br>GSK2269557 Pharmacokinetic Parameters | Parameters with units | SAC [1] |

# 10.8.6. Pharmacokinetic Figures

| Pharma | Pharmacokinetic Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Individ | Individual Concentration Plots | | | | |
| 3.1 | PK | PK16 | Individual GSK2269557 Plasma Concentration-Time Plot by Subject (Linear and Semi-log) | Paginate by Subject | SAC [1] |
| Mean / | Mean / Median Concentration Plots | | | | |
| 3.2 | PK | PK20 | Median (range) Plasma GSK2269557 Concentration-<br>Time Plots (Linear and Semi-log) | Paginate by Treatment | SAC [1] |

# 10.8.7. ICH Listings

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Rando | Randomisation | | | | |
| 1 | Safety | CP_TA1 | Listing of Randomised and Actual Treatments | | SAC [1] |
| Subjec | Subject Disposition | | | | |
| 2 | Safety | ES2 | Listing of Reasons for Study Withdrawal | | SAC [1] |
| 3 | APE | ES7 | Listing of Reasons for Screening Failure | | SAC [1] |
| 4 | Safety | BL1 | Listing of Subjects for Whom the Treatment Blind was Broken | | SAC [1] |
| 5 | Safety | SP3 | Listing of Subjects Excluded from PK Population | | SAC [1] |
| 6 | Safety | DV2 | Listing of Important Protocol Deviations | | SAC [1] |
| 7 | Safety | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC [1] |
| Demog | Demographics | | | | |
| 8 | Safety | DM2 | Listing of Demographic Characteristics | | SAC [1] |
| 9 | Safety | DM9 | Listing of Race | | SAC [1] |
| Prior and Concomitant Medications | | | | | |
| 10 | Safety | CP_CM3 | Listing of Concomitant Medications | | SAC [1] |
| 11 | Safety | MH2 | Listing of Current and/or Past Medical Conditions | | |

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Exposi | Exposure and Treatment Compliance | | | | |
| 12 | Safety | EX3 | Listing of Exposure Data | | SAC [1] |
| Advers | e Events | | | | |
| 13 | Safety | AE7 | Listings of Subject Numbers for Individual Adverse Events | | SAC [1] |
| 14 | Safety | AE8 | Listing of All Adverse Events | | SAC [1] |
| 15 | Safety | AE8 | Listing of Serious Adverse Events | | SAC [1] |
| 16 | Safety | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | | SAC [1] |
| LABS | | | | | |
| 17 | Safety | CP_LB5 | Listing of All Clinical Chemistry Laboratory Data for Subjects with PCI Abnormalities | | SAC [1] |
| 18 | Safety | CP_LB5 | Listing of All Haematology Laboratory Data for Subjects with PCI Abnormalities | | SAC [1] |
| 19 | Safety | CP_LB5 | Listing of Clinical Chemistry Abnormalities of Potential Clinical Importance | | |
| 20 | Safety | CP_LB5 | Listing of Haematology Abnormalities of Potential Clinical Importance | | |
| ECGs | ECGs | | | | |

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 21 | Safety | CP_EG3 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | | SAC [1] |
| 22 | Safety | CP_EG3 | Listing of ECG Values of Potential Clinical Importance | | SAC [1] |
| 23 | Safety | CP_EG5 | Listing Abnormal ECG Findings | | SAC [1] |
| Vital Si | gns | | | | |
| 24 | Safety | CP_VS4 | Listing of All Vital Signs for Subjects with Any Value of Potential Clinical Importance | | SAC [1] |
| 25 | Safety | CP_VS4 | Listing of Vital Signs of Potential Clinical Importance | | SAC [1] |
| Spiron | Spirometry | | | | |
| 26 | Safety | | Listing of Spirometry (FEV1 and FVC) | See example:<br>uk1salx00175/gsk2269557/mid205759/final/<br>Listing 61 | SAC [1] |
| PK | PK | | | | |
| 27 | PK | PK07 | Listing of GSK2269557 Plasma Pharmacokinetic Concentration-Time Data | | SAC [1] |
| 28 | PK | PK13 | Listing of Derived Plasma GSK2269557<br>Pharmacokinetic Parameters | | SAC [1] |